



# PARTICIPANT INFORMATION SHEET

| STUDY TITLE: | |
|---|---|
| "Interventional study focused on pro | oviding personalised health recommendations to the general population |
| through an integrated Alguided app | as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |

We are writing to inform you about a research study in which you are invited to take part in. The study has been approved by the centre's Research Ethics Committee, in accordance with current legislation, Law 14/2007, 3 July on Biomedical Research. Our aim is that you receive sufficient accurate information to make an informed decision on whether or not to participate in this study. Please take the time to read this information sheet carefully. You may contact us at any time to clarify any doubts that may arise. You may also discuss this project with others if you wish. Additionally, you may request further explanations about any aspect of the study and its implications by contacting the project's principal investigator, Name, by telephone on XXXXXXXXXX.

#### 1. Voluntary participation

You have been invited to participate in this study because you require a gastroscopy (a process in which a camera is inserted into your stomach via a scope through your mouth and down your throat) due to a suspected diagnosis of chronic gastric inflammation or because you were previously diagnosed with an infection by the *Helicobacter pylori* bacterium (a bacteria that infections the stomach). You should know that your participation in this study is voluntary and that you may decide NOT to participate. If you decide to participate, you can change your decision and withdraw consent at any time – your choice will not alter your relationship with your doctor or negatively affect the health care you receive. Your acceptance to participate in this study implies your consent to treat some of your personal data, in the manner described below.

# 2. Justification and Objective of the study

This study is carried out to better understand how inflammation over a long period of time may cause changes in the cells that line the stomach (gastric epithelium) and can eventually develop into cancer. Understanding the changes that occur before cancer develops allows for patients at risk to be identified early and to be guided with strict follow-ups as a prevention strategy.

The main objective of this study is to develop a tool that will be assisted by artificial intelligence (AI), and will combine clinical data, risk factors such as Helicobacter pylori infection (a common bacterial infection of the stomach), and pathological and molecular risks of inflammation of the stomach tissue in order to apply more effective prevention measures of gastric cancer, in the future.

#### 3. Description of the study

This study is part of the strategy of the project: "European Consortium for the development of a tool assisted by artificial intelligence for the diagnosis and management of chronic gastric inflammation".

The study will be carried out in 2 parts:

#### First phase

Participating patients will be classified into one of 3 risk levels (high, medium-low), based on their health status, preexisting conditions, history of Helicobacter pylori infection, history of changes in the gastric epithelium, or family history of cancer and will receive health recommendations based on their risk, which will be calculated based on the literature, in order to provide recommendations aligned with the clinical best practice guidelines.



# DEPARTAMENT CLÍNIC MALVA-ROSA

#### **Hospital Clínic Universitari**

A health questionnaire will be completed, and biopsy samples will be collected during the gastroscopy indicated by your treating physician, which will be analysed according to the protocol of the study to complete your individual risk profile.

Your participation will also consist of a dynamic monitoring process where your quality of life and your state of health. Additionally, the *Helicobacter pylori* eradication status (in the event that you received eradication treatment) will be measured to assess if the treatment was effective or not. Adherence to the established guidelines for follow-up in your case will be also monitored.

The expected number of patients to be recruited in this project is 450 patients (150 cases and 150 healthy controls as well as 150 gastric cancer patients to train the system).

#### Second phase

During the second phase of the project, the risk prediction capabilities of the AI-assisted tool will be established and improved, after integrating the data of the patients recruited in the initial phase, the recommendations given to the patient cohort will be reviewed. You will be informed of this update by your attending physician.

This is an international multicentre study in which 9 hospitals across Europe will participate. Participating countries include Spain, Portugal, France, Latvia, Lithuania, and the Netherlands, and recruitment is expected to take place in 3 years.

This study seeks to develop a clinical tool that is useful in the prevention of gastric cancer.

#### 4. Study activities

The entire project will last 4 years.

Your participation, should you agree, will consist of answering questions about your state of health approximately every 2 months throughout the duration of the study, and the analysis of your gastric biopsy samples, with 5 additional biopsies, which would also be performed as part of the diagnosis process. In the event that you participate in the multiomic study (which involves analyzing the samples in greater depth including a molecular study, and analysis of the immune microenvironment and the microbiome), 5 more biopsies will be collected, in addition to two samples of blood (5 mL EDTA tubes— EDTA is an anticoagulant and keeps the blood from clotting), and saliva and fecal samples (see the figure).

Collection of these samples will not involve any modification to your treatment.

The biopsy samples will be sent to I3S (Portugal) for characterization and classification, accompanied by the local pathology report.







In addition, to analyze the influence of exposure to different risk factors between cases, you will be asked simple questions related to your diet, anthropometry (physical measures including weight and height), physical activity, socioeconomic status, tobacco, alcohol, and salt consumption, as well as medical history related to gastritis and your family history of cancer.

The data from your medical history will be included in an electronic database, exclusive to the project, in an encrypted or coded form so that you cannot be directly identified; this will be shared and analyzed by the entire research team. The conclusions will be published and disseminated to the scientific community and the general population.

The data collected will undergo validation processes that will guarantee its integrity, consistency, and reliability.

#### 5. Risks and inconveniences derived from your participation in the study

The risks and discomfort will be those derived from the indicated gastroscopy, a process in which a camera is inserted into your stomach via a scope through your mouth and down your throat. You may have some throat and stomach pain from the gastroscopy, as well as a little bleeding resulting from the biopsies. This is normal and should pass within a few hours. Should it persist, please contact the project's principal investigator.

For most people, needle sticks to draw blood are not a problem. However, on occasion, they can cause bleeding, bruising, discomfort, infection and/or pain at the point of blood extraction. You may also feel dizzy. Should you feel any of these symptoms, please notify the nurse performing the blood draw.

#### 6. Possible benefits

It is very possible that you will not gain any benefit to your health from participating in this study, but it may help to better understand your disease and improve the prognosis and treatment of future patients.

# 7. Protection of personal data

The processing of your personal data related to this study will be carried out in compliance with Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on Data Protection (GDPR). And it is carried out under the co-responsibility of the following institutions:

| Institution | Country | Id. code | Contact |
|---------------------------|----------------|-------------|----------------|
| IIS INCLIVA | Spain | ESG96886080 | www.incliva.es |
| 135 | Portugal | | |
| UniversityofLatvia | Latvia | | |
| Hospital La Princesa | Spain | | |
| Hospital Clinic Barcelona | Spain | | |
| CHU Nantes | France | | |
| LithuaniaUniversity | Lithuania | | |
| Instituto Portugués de | Portugal | | |
| Oncologia | | | |
| Erasmus Medical Center | TheNetherlands | | |

The personal data that this study requires will be taken from questionnaire that you will complete, existing data in your clinical records and the results of the testing you will undergo, which will be included in an electronic database specific to the project, in an encrypted format, without directly identifiable data, for subsequent analysis by the entire research team. The conclusions will be published and disseminated to the scientific community and the general public. Your identity will not be revealed to any person, with the exceptions of medical emergency or legal requirement. This study's data can be transmitted to third parties and to other countries, but in no case containing information that can identify you directly. If data transfer takes place, it will be for the study purposes previously described or for use in scientific





publications, but always maintaining confidentiality and identity protection in accordance with current legislation. Information and updates on the progress of this study can be found on the following website:......

If data obtained in this study may be clinically or genetically relevant to you, and of interest and importance to your health or that of your family, it may be requested that you be informed by your study doctor. In the instance that you should express your refusal to be informed, and in the opinion of the doctor in charge, the information obtained is necessary to avoid serious damage to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting the centre's Ethics Committee. This information will be communicated by professionals who are able to explain its relevance and the options that may be open to you. In case of clinically relevant genetic information, you may receive the necessary genetic counselling.

Although it is unlikely, genetic information may be obtained that is not directly related to the primary objective of the analysis, but that is considered clinically relevant to your health, or that of your family in case of heritable alterations. If so, ask your doctor about the implications of this information. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant for your family members. It is your personal decision to inform them, something we strongly recommend, so that if they wish they may seek further medical advice and guidance at a specialized clinic for family cancer or clinical genetics, where they will be informed about the clinical significance of the identified disorder.

In accordance with data protection legislation, you may exercise your right to access, modify, oppose and cancel data by contacting your study doctor. If you decide to withdraw consent to participate in this study, no new data will be added to the database, but the existing data will be used. Additionally, you can limit the processing of incorrect data, and may request a copy or transfer to a third party (portability) of any data you have provided for the study. To exercise your rights, contact your study doctor or the centre's Data Protection Officer at protectiondatos@incliva.es. Also, please note that if you are not satisfied with the way your request is handled, you have the right to contact the Spanish Data Protection Agency at www.aepd.es/agencia/contacto.

It is quite likely that you will not see any benefit to your health from participating in this study, but it could help you to understand your disease better and improve prognosis and treatment of future patients.

# 8. Information relating to biological samples

Your participation in this study entails obtaining and using biological samples for research purposes, which will be carried out in accordance with the provisions of Law 14/2007 on biomedical research and Royal Decree 1716/2011 on Biobanks, regulations that guarantee the Respect for the rights that assist you.

By signing this document, you agree that your samples will be used for the purposes of this study.

During this study, biopsy samples will be collected during the gastroscopy that will be performed for the diagnosis of your disease, blood, saliva and stools as described in section 4, study activities.

The biological samples will be processed by the different clinical centres included in the table in section 7. And if you allow it, the surplus of biological material will be stored in the IIS INCLIVA Biobank for use in subsequent research projects.

#### 8.1 Sample Collection Procedures, Discomfort, and Potential Risks

The samples will be obtained as described in section 4, titled Study activities and obtaining them could cause you the inconvenience described in section 5, titled Risks and inconveniences derived from your participation in the study.

The samples will be associated with a code that can only be related to their identity by authorized personnel, in the same way that has been previously explained with the data obtained during the study.

The data derived from the use of these samples will be treated in the same way as the rest of the data obtained during this study in terms of data protection.





The samples and associated data will be kept under adequate security conditions, and it is guaranteed that the subjects cannot be identified through means considered reasonable by persons other than those authorized.

Some additional data or samples may be required. In this case, your doctor will contact you to request your collaboration again. You will be informed of the reasons and your consent will be requested again.

#### 8.2 Expected benefits

You will not receive any economic benefit from the donation of the samples and the transfer of the data provided, nor will you have rights to possible commercial benefits of the discoveries that may be achieved because of the research carried out.

#### 8.3. Place of analysis and storage of samples

The study biopsy samples will be sent to I3s (Portugal). I3s will distribute part of the samples to CHU Nantes and the University of Lithuania to jointly carry out the necessary determinations for the study.

#### 8.4. Implications of the information obtained when analysing the samples

If you request it, you may be provided with information about the general objectives of this study.

If this study obtains data that could be clinically or genetically relevant to you, and of interest to your health or that of your family, you may request that they be communicated to you by your study doctor.

In the instance that you should express your refusal to be informed, and according to the criteria of the responsible doctor, the information obtained is necessary to avoid serious harm to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting to the Healthcare Ethics Committee of the centre. The communication of this information will be carried out by professionals who are able to adequately explain its relevance and the options that could be considered. In the case of clinically relevant genetic information, you may receive the mandatory genetic counselling.

Although unlikely, genetic information obtained that is not directly related to the primary objective of the analysis, may be considered clinically relevant to your health, or that of your family in case of heritable disorders. If so, discuss the implications of this information with your doctor. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant to your biological relatives. It is your personal decision to inform them, something that we recommend, so that if they so wish, they can seek out a specialized consultation in family cancer or clinical genetics, where they will be informed about the clinical significance of the identified alteration.

#### 8.5. Future use of samples

Once the study is finished, the remaining samples will be destroyed, unless you consent to storage in a Biobank regime to be used in future research. In this case, the samples will be stored in the INCLIVA Biobank. From there they will be transferred for projects provided there is a favourable opinion from the scientific committee and the Ethics committee of the Biobank.

You can contact the INCLIVA biobank to biobanco@incliva.es to obtain information on the projects in which your samples have been used.

Said authorization can be granted by signing the corresponding consent of the INCLIVA Biobank. If you change your mind, you have the right to request its destruction or anonymization, this can be done through your study doctor or through direct communication to the biobank. However, it is important that you understand that the data obtained in the analyses carried out up to that moment may be used for the requested purposes and may be kept in compliance with the corresponding legal obligations.

Should you request it, the biobank will provide you with information about the research projects in which your samples have been used.





# INFORMED CONSENT

| INFORIVIED CONSENT | |
|---|---|
| STUDY TITLE: | |
| • | on providing personalised health recommendations to the general population |
| | d app as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |
| I. | < <participant's and="" name="" surname="">&gt;</participant's> |
| (Name in handwriting by the | e patient) |
| have read the information sheet t | hat has been given to me about the study. |
| I was able to ask questions about | • |
| I have received enough information | |
| I have spoken to | < <name investigator="" of="">&gt; in handwriting by the patient)</name> |
| I understand that my participation | |
| I understand that I am free to witl | |
| - At any time. | |
| - Without giving a reason. | |
| - Without this affecting my medic | al care. |
| I freely give my consent to particip | pate in the study. |
| I consent to the use and processing | ng of my personal data for this investigation under the conditions explained in |
| this information sheet. | |
| <u>Use of Samples</u> | |
| I consent to the storage and use | e of the samples and associated data for this research under the conditions |
| explained in this information shee | · |
| • | |
| □YES □NO | |
| I would like the study doctor to | inform me about information generated from the research (genetic or non- |
| | hat may be relevant and applicable to my health or that of my family members: |
| □YES □NO | Contact telephone or email |
| | · |
| I consent to be contacted if there | is a need for further information or additional biological samples. |
| □YES □NO | Contact telephone or email |
| I will receive a signed and dated c | opy of this informed consent form |
| i wiii receive a signed and dated c | opy of this informed consent form |
| Participant's Signature | Investigator's Signature |
| Date:/ | Date:/ |
| (Signature and date in handwriting by | patient) |







# INFORMED CONSENT LEGALREPRESENTATIVE

| through an integrated Alguided ar | providing personalised health recommendations to the general population<br>op as a strategy for gastric cancer prevention". |
|---|---|
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |
| ,(Name in handwriting by represon my capacity as | <pre> &lt;<representative's and="" name="" surname="">&gt; entative)</representative's></pre> |
| <u></u> | <pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;</pre></pre></pre></pre> <pre></pre> |
| (Name in handwriting by repres | |
| was able to ask questions about the have received enough information a have spoken to | <pre>chout the study&lt;<name investigator="" of="">&gt; andwriting by representative) n is voluntary.</name></pre> |
| n this information sheet. | |
| Use of Samples consent to the storage and use of explained in this information sheet. | the samples and associated data for this research under the condition |
| YES NO | |
| would like the study doctor to inf<br>genetic, depending on the case) that | orm me about information generated from the research (genetic or nor may be relevant and applicable to my health or that of my family members Contact telephone or email |
| would like the study doctor to infgenetic, depending on the case) that<br>YES<br>NO | may be relevant and applicable to my health or that of my family members |
| would like the study doctor to inf<br>genetic, depending on the case) that<br>YES NO<br>consent to be contacted if there is a | may be relevant and applicable to my health or that of my family members Contact telephone or email need for further information or additional biological samples. Contact telephone or email |
| would like the study doctor to infigenetic, depending on the case) that YES NO consent to be contacted if there is a YES NO | may be relevant and applicable to my health or that of my family members Contact telephone or email need for further information or additional biological samples. Contact telephone or email of this informed consent form |







# INFORMED CONSENT BEFORE WITNESSES

| STUDY TITLE: | |
|---|---|
| "Interventional study focused or | n providing personalised health recommendations to the general population |
| through an integrated Alguided a | app as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |
| l, | < <witness's and="" name="" surname="">&gt;</witness's> |
| (Name in handwriting by with | |
| as a witness, state that in my prese | |
| | (Name in handwriting by witness) |
| has been informed and has read | I the information sheet about the study, and therefore: |
| | <i>,</i> , |
| He/she has read the information sh | neet that has been given to him/her about the study. |
| Was able to ask questions about the | · |
| Has received enough information a | bout the study. |
| Has spoken to | |
| • | handwriting by witness) |
| Understands that his/her participat | · |
| Understands that he/she is free to | withdraw from the study: |
| - At any time. | |
| - Without giving a reason. | |
| - Without this affecting his/her med | |
| Freely gives his/her consent to part | · |
| _ | of his/her personal data for this investigation under the conditions explained |
| in this information sheet. | |
| <u>Use of Samples</u> | |
| Constant to the standard section | of the considerated and the delegation of the constant of the |
| | of the samples and associated data for this research under the conditions |
| explained in this information sheet. | |
| □YES □NO | |
| Mould like the study deeter to infe | arm him/har about information gonerated from the research (gonetic or non |
| • | orm him/her about information generated from the research (genetic or non- |
| | at may be relevant and applicable to his/her health or that of his/her family |
| members: | |
| □YES □NO | Contact telephone or email |
| Consents to be contacted if there is | a a need for further information or additional biological camples |
| | s a need for further information or additional biological samples. |
| YES NO | Contact telephone or email |
| Will receive a signed and dated cop | ay of this informed consent form |
| will receive a signed and dated cop | y or this informed consent form |
| Signature of witness | Investigator's Signature |
| Date:/ | Date:/ |
| (Signature and date in handwriting by v | |





# **PARTICIPANT INFORMATION SHEET**

| STUDY TITLE: | |
|---|---|
| "Interventional study focused on pro | oviding personalised health recommendations to the general population |
| through an integrated AI guided app | as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |

#### 1. Voluntary participation

You have been invited to participate in this study because you have been diagnosed with gastric cancer and you will undergo an endoscopy, as a strategy for managing your disease. By agreeing to participate in this study you grant us your consent to access and process some of your personal data in the ways described below, and to take extra biopsies or samples of the tissue from the gastric mucosa which makes up the inner lining of the stomach, and also to collect of a sample of blood (2 EDTA tubes 5 mL each – EDTA is an anticoagulant and keeps the blood from clotting), saliva and faecal samples. Collection of these samples will not involve any modification to your treatment. You should know that your participation in this study is voluntary and that you can decide NOT to participate. If you decide to participate, you may change your mind and withdraw your consent at any time- your choice will not affect your relationship with your doctor or negatively affect the health care you receive.

#### 2. Justification and Objective of the study

This study is carried out to better understand how inflammation over a long period of time may cause changes in the cells that line the stomach (gastric epithelium) and can eventually develop into cancer. Understanding the changes that occur before cancer develops allows for patients at risk to be identified early and to be guided with strict follow-ups as a prevention strategy.

The main objective of this study is to develop a tool that will be assisted by artificial intelligence (AI), and will combine clinical data, risk factors such as *Helicobacter pylori* infection (a common bacterial infection of the stomach), and pathological and molecular risks of inflammation of the stomach tissue in order to apply more effective prevention measures of gastric cancer, in the future.

#### 3. Description of the study

This study is part of the strategy of the project: "European Consortium for the development of a tool-assisted by artificial intelligence for the diagnosis and management of chronic gastric inflammation".

A health questionnaire will be completed, and biopsy samples will be collected during the gastroscopy indicated by your treating physician, your participation will allow the project to develop the AI-assisted tool.

The expected number of patients to be recruited in this project is 450 patients (150 cases, 150 controls 150 gastric cancer controls to train the system).





This is an international multicentre study in which 9 hospitals in Europe will participate. Participating countries include Spain, Portugal, France, Latvia, Lithuania, and the Netherlands, and recruitment is expected to take place in 3 years.

This study seeks to develop a clinical tool that is useful in the prevention of gastric cancer.

#### 4. Study activities

The entire project will last 4 years.

Your participation, should you agree, will consist of the analysis of your gastric biopsy samples, 5 additional biopsies, two samples of blood (5 mL EDTA tubes), saliva and fecal collection (see the figure). It will not imply any modification of your treatment.

The biopsy samples will be sent to I3S (Portugal) for characterization and classification, accompanied by the local pathology report.



In addition, to analyze the influence of exposure to different risk factors between cases, you will be asked simple questions related to your diet, anthropometry (physical measures including weight and height), physical activity, socioeconomic status, tobacco, alcohol, and salt consumption, as well as medical history related to gastritis and your family history of cancer.

The data from your medical history will be included in an electronic database, exclusive to the project, in an encrypted or coded form so that you cannot be directly identified; this will be shared and analyzed by the entire research team. The conclusions will be published and disseminated to the scientific community and the general population.

The data collected will undergo validation processes that will guarantee its integrity, consistency, and reliability.

#### 5. Risks and inconveniences derived from your participation in the study

The risks and discomfort will be those derived from the indicated gastroscopy, a process in which a camera is inserted into your stomach via a scope through your mouth and down your throat. You may have some throat and stomach pain from the gastroscopy, as well as a little bleeding resulting from the biopsies. This is normal and should pass within a few hours. Should it persist, please contact the project's principal investigator.

For most people, needle sticks to draw blood are not a problem. However, on occasion, they can cause bleeding, bruising, discomfort, infection and/or pain at the point of blood extraction. You may also feel dizzy. Should you feel any of these symptoms, please notify the nurse performing the blood draw.





#### 6. Possible benefits

It is very possible that you will not gain any benefit to your health from participating in this study, but it may help to better understand your disease and improve the prognosis and treatment of future patients.

#### 7. Protection of personal data

The processing of your personal data related to this study will be carried out in compliance with Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on Data Protection (GDPR). And it is carried out under the co-responsibility of the following institutions:

| Institution | Country | Id. code | Contact |
|---|---|---|---|
| IIS INCLIVA | Spain | ESG96886080 | www.incliva.es |
| 13S | Portugal | | |
| University of Latvia | Latvia | | |
| Hospital La Princesa | Spain | | |
| Hospital Clinic Barcelona | Spain | | |
| CHU Nantes | France | | |
| Lithuania University | Lithuania | | |
| Instituto Portugués de Oncologia | Portugal | | |
| Erasmus Medical Center | TheNetherlands | _ | |

Your identity will not be revealed to any person, with the exceptions of medical emergency or legal requirements. This study's data can be transmitted to third parties and to other countries, but in no case containing information that can identify you directly. If data transfer takes place, it will be for the study purposes previously described or for use in scientific publications, but always maintaining confidentiality and identity protection in accordance with current legislation. Information and updates on the progress of this study can be found on the following website:......

If data obtained in this study may be clinically or genetically relevant to you, and of interest and importance to your health or that of your family, it may be requested that you be informed by your study doctor. In the instance that you should express your refusal to be informed, and in the opinion of the doctor in charge, the information obtained is necessary to avoid serious damage to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting the centre's Ethics Committee. This information will be communicated by professionals who are able to explain its relevance and the options that may be open to you. In case of clinically relevant genetic information, you may receive the necessary genetic counselling.

Although it is unlikely, genetic information may be obtained that is not directly related to the primary objective of the analysis, but that is considered clinically relevant to your health, or that of your family in case of heritable alterations. If so, ask your doctor about the implications of this information. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant for your family members. It is your personal decision to inform them, something we strongly recommend, so that if they wish they may seek further medical advice and guidance at a specialized clinic for family cancer or clinical genetics, where they will be informed about the clinical significance of the identified disorder.

In accordance with data protection legislation, you may exercise your right to access, modify, oppose and cancel data by contacting your study doctor. If you decide to withdraw consent to participate in this study, no new data will be added to the database, but the existing data will be used. Additionally, you can limit the processing of incorrect data, and may request a copy or transfer to a third party (portability) of any data you have provided for the study. To exercise your rights, contact your study doctor or the centres Data Protection Officer at <a href="mailto:protectiondatos@incliva.es">at protectiondatos@incliva.es</a>. Also, please note that if you are not satisfied with the way your request is handled, you have the right to contact the <a href="mailto:Spanish">Spanish</a> Data Protection Agency at <a href="mailto:www.aepd.es/agencia/contacto">www.aepd.es/agencia/contacto</a>.

It is quite likely that you will not see any benefit to your health from participating in this study, but it could help you to understand your disease better and improve prognosis and treatment of future patients.





#### 8. Information relating to biological samples

Your participation in this study entails obtaining and using biological samples for research purposes, which will be carried out in accordance with the provisions of Law 14/2007 on biomedical research and Royal Decree 1716/2011 on Biobanks, regulations that guarantee the Respect for the rights that assist you.

By signing this document, you agree that your samples will be used for the purposes of this study.

During this study, biopsy samples will be collected during the gastroscopy that will be performed for the diagnosis of your disease, blood and saliva as described in section 4, study activities.

The biological samples will be processed by the different clinical centres included in the table in section 7. And if you allow it, the surplus of biological material will be stored in the IIS INCLIVA Biobank for use in subsequent research projects.

#### 8.1 Sample Collection Procedures, Discomfort, and Potential Risks

The samples will be obtained as described in section 4, titled Study activities and obtaining them could cause you the inconvenience described in section 5, titled Risks and inconveniences derived from your participation in the study.

The samples will be associated with a code that can only be related to their identity by authorized personnel, in the same way that has been previously explained with the data obtained during the study.

The data derived from the use of these samples will be treated in the same way as the rest of the data obtained during this study in terms of data protection.

The samples and associated data will be kept under adequate security conditions, and it is guaranteed that the subjects cannot be identified through means considered reasonable by persons other than those authorized.

Some additional data or samples may be required. In this case, your doctor will contact you to request your collaboration again. You will be informed of the reasons and your consent will be requested again.

#### 8.2 Expected benefits

You will not receive any economic benefit from the donation of the samples and the transfer of the data provided, nor will you have rights to possible commercial benefits of the discoveries that may be achieved because of the research carried out.

#### 8.3. Place of analysis and storage of samples

The study biopsy samples will be sent to I3s (Portugal). I3s will distribute part of the samples to CHU Nantes and the University of Lithuania to jointly carry out the necessary determinations for the study.

#### 8.4. Implications of the information obtained when analysing the samples

If you request, you may be provided with information about the general studies of this study.

If this study obtains data that could be clinically or genetically relevant to you, and of interest to your health or that of your family, you may request that they be communicated to you by your study doctor.

In the instance that you should express your refusal to be informed, and according to the criteria of the responsible doctor, the information obtained is necessary to avoid serious harm to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting to the Healthcare Ethics Committee of the centre. The communication of this information will be carried out by professionals who are able to adequately explain its relevance and the options that could be considered. In the case of clinically relevant genetic information, you may receive mandatory genetic counselling.





Although unlikely, genetic information obtained that is not directly related to the primary objective of the analysis, may be considered clinically relevant to your health, or that of your family in case of heritable disorders. If so, discuss the implications of this information with your doctor. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant to your biological relatives. It is your personal decision to inform them, something that we strongly recommend, so that if they so wish, they can seek out a specialized consultation in family cancer or clinical genetics, where they will be informed about the clinical significance of the identified alteration.

#### 8.5. Future use of samples

Once the study is finished, the remaining samples will be destroyed, unless you consent to storage in a Biobank regime to be used in future research. In this case, the samples will be stored in the INCLIVA Biobank. From there they will be transferred for projects provided there is a favourable opinion from the scientific committee and the Ethics committee of the Biobank.

You can contact the INCLIVA biobank to biobanco@incliva.es to obtain information on the projects in which your samples have been used.

Said authorization can be granted by signing the corresponding consent of the INCLIVA Biobank. If you change your mind, you have the right to request its destruction or anonymization, this can be done through your study doctor or through direct communication with the biobank. However, it is important that you understand that the data obtained in the analyses carried out up to that moment may be used for the requested purposes and may be kept in compliance with the corresponding legal obligations.

Should you request it, the biobank will provide you with information about the research projects in which your samples have been used.







# **INFORMED CONSENT**

| STUDY TITLE: | |
|---|---|
| "Interventional study focused on pro | oviding personalised health recommendations to the general population |
| through an integrated AI guided app | as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |

| l, | | < <pa< th=""><th>articipant's name and surname&gt;&gt;</th><th></th></pa<> | articipant's name and surname>> | |
|---|---|---|---|---|
| (Name in | handwriting by the patient | | | |
| have read the info | rmation sheet that has | been given to me abou | out the study. | |
| I was able to ask qu | uestions about the stu | dy. | | |
| I have received end | ough information abou | t the study. | | |
| I have spoken to _ | (Name in handw | | <pre>&lt;<name investigator="" of="">&gt;</name></pre> | |
| | my participation is volu | | | |
| | am free to withdraw f | rom the study: | | |
| - At any time. | | | | |
| - Without giving a | | | | |
| - Without this affect | cting my medical care. | | | |
| | nsent to participate in | - | | |
| | | y personal data for this | is investigation under the conditions explained | in |
| this information sh | ieet. | | | |
| Use of Samples | | | | |
| I consent to the s explained in this in | | e samples and associat | ated data for this research under the condition | ons |
| YYES | Ϋ́NO | | | |
| | • | be relevant and applic | on generated from the research (genetic or no icable to my health or that of my family member or email | |
| I consent to be cor | ntacted if there is a nee | ed for further information | tion or additional biological samples. | |
| YYES | Ϋ́NO | Contact telephone o | or email | |
| I will receive a sign | ed and dated copy of t | his informed consent fo | form | |
| 223 2 2 3 3 5 1 | 200 200, 01 | | | |
| Participant's Sig | | Dat | vestigator's Signature<br>ate:/ | |







# INFORMED CONSENT LEGAL REPRESENTATIVE

| | providing personalised health recommendations to the general population |
|---|---|
| STUDY CODE | op as a strategy for gastric cancer prevention". 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |
| <u> </u> | |
| l, | <pre>&lt;<representative's and="" name="" surname="">&gt;</representative's></pre> |
| (Name in handwriting by represen | |
| In my capacity as | <pre> &lt;<relationship participant="" the="" to="">&gt;, of</relationship></pre> <pre></pre> <pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre></pre><pre>&lt;</pre></pre> |
| (Name in handwriting by represen | |
| have read the information sheet that h | |
| I was able to ask questions about the st | · |
| I have received enough information about have spaken to | |
| I have spoken to(Name in hand | dwriting by representative) |
| I understand that his/her participation | |
| I understand that he/she is free to with | · |
| - At any time. | , |
| - Without giving a reason. | |
| - Without this affecting his/her medical | l care. |
| I freely give my consent to his/her part | |
| | nis/her personal data for this investigation under the conditions explained |
| in this information sheet. | |
| Use of Samples | |
| I consent to the storage and use of t | he complete and acceptated data for this research under the conditions |
| explained in this information sheet. | the samples and associated data for this research under the conditions |
| • | |
| Yyes Yno | |
| • | m me about information generated from the research (genetic or non-<br>ay be relevant and applicable to my health or that of my family members: |
| Yyes Yno | Contact telephone or email |
| I consent to be contacted if there is a n | eed for further information or additional biological samples. |
| YYES YNO | Contact telephone or email |
| 11125 | Contact telephone of email |
| I will receive a signed and dated copy o | f this informed consent form |
| Signature of legal representative, re | lative or related Investigator's Signature |
| party<br>Date: / / | Date: / / |
| Date. / / | Date. / / |

(Signature and date in handwriting by representative)







# **INFORMED CONSENT BEFORE WITNESSES**

| | STUDY CODE | app as a strategy for gastric cancer prevention". 101095359 – AIDA |
|---|---|---|
| | PRINCIPAL INVESTIGATORS | To be completed |
| | DEPARTMENT | To be completed |
| | CENTER | To be completed |
| l, _ | | < <wirtness's and="" name="" surname="">&gt;</wirtness's> |
| 20 | (Name in handwriting by witness a witness, state that in my presence | |
| us | a withess, state that in my present | (Name in handwriting by witness) |
| ۵ | | ne information sheet about the study, and therefore: |
| | as able to ask questions about the s | , |
| | s received enough information abo | , |
| | s spoken to | <pre></pre> <pre></pre> <pre></pre> <pre></pre> |
| | • | ndwriting by witness) |
| | derstands that his/her participation derstands that he/she is free to wi | · |
| | t any time. | thuraw from the study. |
| | Vithout giving a reason. | |
| | Vithout this affecting his/her medic | al care. |
| | eely gives his/her consent to partici | |
| | • | f his/her personal data for this investigation under the conditions explained |
| in t | this information sheet. | |
| Us | e of Samples | |
| | nsent to the storage and use of plained in this information sheet. | the samples and associated data for this research under the conditions |
| $\Upsilon_{Y}$ | yes Yno | |
| gei | · | n him/her about information generated from the research (genetic or non-may be relevant and applicable to his/her health or that of his/her family |
| Υ | yes Yno | Contact telephone or email |
| Со | nsents to be contacted if there is a | need for further information or additional biological samples. |
| | yes Yno | Contact telephone or email |
| Wi | II receive a signed and dated copy | of this informed consent form |
| | Signature of witness | Investigator's Signature |

Date: \_\_\_\_/\_\_\_\_

Date: \_\_\_/\_\_/\_\_(Signature and date in handwriting by witness)





# PARTICIPANT INFORMATION SHEET

| STUDY TITLE: | |
|---|---|
| "Interventional study focused on pr | oviding personalised health recommendations to the general population |
| through an integrated AI guided app | as a strategy for gastric cancer prevention". |
| STUDY CODE | 101095359 – AIDA |
| PRINCIPAL INVESTIGATORS | To be completed |
| DEPARTMENT | To be completed |
| CENTER | To be completed |

We are writing to inform you about a research study in which you are invited to take part in. The study has been approved by the centre's Research Ethics Committee, in accordance with current legislation, Law 14/2007, 3 July on Biomedical Research. Our aim is that you receive sufficient accurate information to make an informed decision on whether or not to participate in this study. Please take the time to read this information sheet carefully. You may contact us at any time to clarify any doubts that may arise. You may also discuss this project with others if you wish. Additionally, you may request further explanations about any aspect of the study and its implications by contacting the project's principal investigator, Name, by telephone on XXXXXXXXXX.

# 1. Voluntary participation

You have been invited to participate in the study because you require a gastroscopy (a process in which a camera is inserted into your stomach via a scope through your mouth and down your throat) for diagnosis purposes and because your profile meets the healthy control criteria for the disease under study. By agreeing to participate in this study you consent for us to access and process some of your personal data in the ways described below. As well as, extra biopsies from gastric mucosa (tissue from the stomach lining), in addition to – blood, saliva and faecal samples.

Collection of these samples will not involve any modification to your treatment.

You should know that your participation in this study is voluntary and that you may decide NOT to participate. If you decide to participate, you can change your decision and withdraw consent at any time – your choice will not alter your relationship with your doctor or negatively affect the health care you receive. Your acceptance to participate in this study implies your consent to treat some of your personal data, in the manner described below.

#### 2. Justification and Objective of the study

This study is carried out to better understand how inflammation over a long period of time may cause changes in the cells that line the stomach (gastric epithelium) and can eventually develop into cancer. Understanding the changes that occur before cancer develops allows for patients at risk to be identified early and to be guided with strict follow-ups as a prevention strategy.

The main objective of this study is to develop a tool that will be assisted by artificial intelligence (AI), and will combine clinical data, risk factors such as Helicobacter pylori infection (a common bacterial infection of the stomach), and pathological and molecular risks of inflammation of the stomach tissue in order to apply more effective prevention measures of gastric cancer, in the future.

# 3. Description of the study

This study is part of the strategy of the project: "European Consortium for the development of a tool assisted by artificial intelligence for the diagnosis and management of chronic gastric inflammation".

The study will be carried out in 2 parts:

#### First phase



# DEPARTAMENT CLÍNIC MALVA-ROSA

#### **Hospital Clínic Universitari**

Participating patients will be classified into one of 3 risk levels (high, medium-low), based on their health status, preexisting conditions, history of Helicobacter pylori infection, history of changes in the gastric epithelium, or family history of cancer and will receive health recommendations based on their risk, which will be calculated based on the literature, in order to provide recommendations aligned with the clinical best practice guidelines.

A health questionnaire will be completed, and biopsy samples will be collected during the gastroscopy indicated by your treating physician, which will be analysed according to the protocol of the study to complete your individual risk profile.

The expected number of patients to be recruited in this project is 450 patients (150 cases, 150 healthy controls and also 150 cancer controls).

### Second phase

During the second phase of the project, the risk prediction capabilities of the AI-assisted tool will be established and improved, after integrating the data of the patients recruited in the initial phase, the recommendations given to the patient cohort will be reviewed. You will be informed on to this update by your attending physician.

This is an international multicentre study in which 9 hospitals across Europe will participate. Participating countries include Spain, Portugal, France, Latvia, Lithuania, and the Netherlands, and recruitment is expected to take place in 3 years.

This study seeks to develop a clinical tool that is useful in the prevention of gastric cancer.

#### 4. Study activities

The project will last 4 years.

Your participation, should you agree, will consist of answering questions about your state of health approximately every 2 months throughout the duration of the study, and the analysis of your gastric biopsy samples, with 5 additional biopsies, which would also be performed as part of the diagnosis process. In the event that you participate in the multiomic study (which involves analyzing the samples in greater depth including a molecular study, and the analysis of the immune microenvironment and the microbiome), 5 more biopsies will be collected, as well as the collection of two samples of blood (5 mL EDTA tubes— EDTA is an anticoagulant and keeps the blood from clotting), and saliva and fecal samples. Collection of these samples will not involve any modification to your treatment.

The biopsy samples will be sent to I3S (Portugal) for characterization and classification, accompanied by the local pathology report.



In addition, to analyze the influence of exposure to different risk factors between cases, you will be asked simple questions related to your diet, anthropometry (physical measures including weight and height), physical activity,





socioeconomic status, tobacco, alcohol, and salt consumption, as well as medical history related to gastritis and your family history of cancer.

The data from your medical history will be included in an electronic database, exclusive to the project, in an encrypted or coded form so that you cannot be directly identified; this will be shared and analyzed by the entire research team. The conclusions will be published and disseminated to the scientific community and the general population.

The data collected will undergo validation processes that will guarantee its integrity, consistency, and reliability.

#### 5. Risks and inconveniences derived from your participation in the study

The risks and discomfort will be those derived from the indicated gastroscopy, a process in which a camera is inserted into your stomach via a scope through your mouth and down your throat. You may have some throat and stomach pain from the gastroscopy, as well as a little bleeding resulting from the biopsies. This is normal and should pass within a few hours. Should it persist, please contact the project's principal investigator.

For most people, needle sticks to draw blood are not a problem. However, on occasion, they can cause bleeding, bruising, discomfort, infection and/or pain at the point of blood extraction. You may also feel dizzy. Should you feel any of these symptoms, please notify the nurse performing the blood draw.

#### 6. Possible benefits

It is very possible that you will not gain any benefit to your health from participating in this study, but it may help to better understand your disease and improve the prognosis and treatment of future patients.

#### 7. Protection of personal data

The processing of your personal data related to this study will be carried out in compliance with Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on Data Protection (GDPR). And it is carried out under the co-responsibility of the following institutions:

| Institution | Country | Id. code | Contact |
|---------------------------|----------------|-------------|----------------|
| IIS INCLIVA | Spain | ESG96886080 | www.incliva.es |
| I3S | Portugal | | |
| UniversityofLatvia | Latvia | | |
| Hospital La Princesa | Spain | | |
| Hospital Clinic Barcelona | Spain | | |
| CHU Nantes | France | | |
| LithuaniaUniversity | Lithuania | | |
| Instituto Portugués de | Portugal | | |
| Oncologia | | | |
| Erasmus Medical Center | TheNetherlands | | |



# DEPARTAMENT CLÍNIC MALVA-ROSA

#### Hospital Clínic Universitari

If data obtained in this study may be clinically or genetically relevant to you, and of interest and importance to your health or that of your family, it may be requested that you be informed by your study doctor. In the instance that you should express your refusal to be informed, and in the opinion of the doctor in charge the information obtained is necessary to avoid serious damage to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting the centre's Ethics Committee. This information will be communicated by professionals who are able to explain its relevance and the options that may be open to you. In case of clinically relevant genetic information, you may receive the necessary genetic counselling.

Although it is unlikely, genetic information may be obtained that is not directly related to the primary objective of the analysis, but that is considered clinically relevant to your health, or that of your family in case of heritable alterations. If so, ask your doctor about the implications of this information. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant for your family members. It is your personal decision to inform them, something we strongly recommend, so that if they wish they may seek further medical advice and guidance at a specialized clinic for family cancer or clinical genetics, where they will be informed about the clinical significance of the identified disorder.

In accordance with data protection legislation, you may exercise your right to access, modify, oppose and cancel data by contacting your study doctor. If you decide to withdraw consent to participate in this study, no new data will be added to the database, but the existing data will be used. Additionally, you can limit the processing of incorrect data, and may request a copy or transfer to a third party (portability) of any data you have provided for the study. To exercise your rights, contact your study doctor or the centre's Data Protection Officer at protecciondatos@incliva.es. Also, please note that if you are not satisfied with the way your request is handled, you have the right to contact the Spanish Data Protection Agency at <a href="https://www.aepd.es/agencia/contacto">www.aepd.es/agencia/contacto</a>.

It is quite likely that you will not see any benefit to your health from participating in this study, but it could help you to understand your disease better and improve prognosis and treatment of future patients.

# 8. Information relating to biological samples

Your participation in this study entails obtaining and using biological samples for research purposes, which will be carried out in accordance with the provisions of Law 14/2007 on biomedical research and Royal Decree 1716/2011 on Biobanks, regulations that guarantee the Respect for the rights that assist you.

By signing this document, you agree that your samples will be used for the purposes of this study.

During this study, biopsy samples will be collected during the gastroscopy that will be performed for the diagnosis of your disease, blood, saliva, and stools as described in section 4, study activities.

The biological samples will be processed by the different clinical centres included in the table in section 7. And if you allow it, the surplus of biological material will be stored in the IIS INCLIVA Biobank for use in subsequent research projects.

#### 8.1 Sample Collection Procedures, Discomfort, and Potential Risks

The samples will be obtained as described in section 4, titled Study activities and obtaining them could cause you the inconvenience described in section 5, titled Risks and inconveniences derived from your participation in the study.

The samples will be associated with a code that can only be related to their identity by authorized personnel, in the same way that has been previously explained with the data obtained during the study.

The data derived from the use of these samples will be treated in the same way as the rest of the data obtained during this study in terms of data protection.

The samples and associated data will be kept under adequate security conditions, and it is guaranteed that the subjects cannot be identified through means considered reasonable by persons other than those authorized.





Some additional data or samples may be required. In this case, your doctor will contact you to request your collaboration again. You will be informed of the reasons and your consent will be requested again.

#### 8.2 Expected benefits

You will not receive any economic benefit from the donation of the samples and the transfer of the data provided, nor will you have rights to possible commercial benefits of the discoveries that may be achieved because of the research carried out.

#### 8.3. Place of analysis and storage of samples

The study biopsy samples will be sent to I3s (Portugal). I3s will distribute part of the samples to CHU Nantes and the University of Lithuania to jointly carry out the necessary determinations for the study.

#### 8.4. Implications of the information obtained when analysing the samples

If you request it, you may be provided with information about the general objectives of this study.

If this study obtains data that could be clinically or genetically relevant to you, and of interest to your health or that of your family, you may request that they be communicated to you by your study doctor.

In the instance that you should express your refusal to be informed, and according to the criteria of the responsible doctor, the information obtained is necessary to avoid serious harm to your health or that of your biological relatives, a close relative or a representative will be informed, after consulting to the Healthcare Ethics Committee of the center. The communication of this information will be carried out by professionals who are able to adequately explain its relevance and the options that could be considered. In the case of clinically relevant genetic information, you may receive the mandatory genetic counselling.

Although unlikely, genetic information obtained that is not directly related to the primary objective of the analysis, may be considered clinically relevant to your health, or that of your family in case of heritable disorders. If so, discuss the implications of this information with your doctor. In case you prefer not to be informed, your decision will be respected. The information obtained may also be relevant to your biological relatives. It is your personal decision to inform them, something that we recommend, so that if they so wish, they can seek out a specialized consultation in family cancer or clinical genetics, where they will be informed about the clinical significance of the identified alteration.

#### 8.5. Future use of samples

Once the study is finished, the remaining samples will be destroyed, unless you consent to storage in a Biobank regime to be used in future research. In this case, the samples will be stored in the INCLIVA Biobank. From there they will be transferred for projects provided there is a favourable opinion from the scientific committee and the Ethics committee of the Biobank.

You can contact the INCLIVA biobank to biobanco@incliva.es to obtain information on the projects in which your samples have been used.

Said authorization can be granted by signing the corresponding consent of the INCLIVA Biobank. If you change your mind, you have the right to request its destruction or anonymization, this can be done through your study doctor or through direct communication to the biobank. However, it is important that you understand that the data obtained in the analyses carried out up to that moment may be used for the requested purposes and may be kept in compliance with the corresponding legal obligations.

Should you request it, the biobank will provide you with information about the research projects in which your samples have been used.





# INFORMED CONSENT

| STUDY TITLE: | | |
|---|---|---|
| | on providing personalised health recommendations to the | general population |
| | d app as a strategy for gastric cancer prevention". | |
| STUDY CODE | 101095359 – AIDA | |
| PRINCIPAL INVESTIGATORS | To be completed | |
| DEPARTMENT | To be completed | |
| CENTER | To be completed | |
| 1 | <pre><pre>&lt;<pre>&lt;<pre></pre></pre></pre></pre> | >> |
| (Name in handwriting by the p | patient) | |
| | at has been given to me about the study. | |
| I was able to ask questions about th | e study. | |
| I have received enough information | | |
| I have spoken to | < <name investiga<="" of="" td=""><td>tor&gt;&gt;</td></name> | tor>> |
| • | handwriting by the patient) | |
| I understand that my participation is<br>I understand that I am free to withd | · | |
| | raw from the study: | |
| <ul><li>At any time.</li><li>Without giving a reason.</li></ul> | | |
| - Without this affecting my medical | caro | |
| I freely give my consent to participa | | |
| | of my personal data for this investigation under the cond | litians avalained in |
| this information sheet. | of my personal data for this investigation under the cond | illions explained in |
| this information sheet. | | |
| Use of Samples | | |
| <u> </u> | | |
| I consent to the storage and use of | of the samples and associated data for this research un | der the conditions |
| explained in this information sheet. | | |
| □YES □NO | | |
| I was la lika tha atualy daatay ta iy | forms are about information concreted from the recent | ah /aanatia au nan |
| · | form me about information generated from the researd<br>t may be relevant and applicable to my health or that of m | |
| □YES □NO | Contact telephone or email | |
| I consent to be contacted if there is | a need for further information or additional biological san | nnles |
| | | • |
| □YES □NO | Contact telephone or email | |
| I will receive a signed and dated cop | y or this informed consent form | |
| Doublein out o Circustore | lancation to de Cinnature | |
| Participant's Signature | Investigator's Signature | |
| Date://(Signature and date in handwriting by page 5.5. | Date:/ | |
| 10.011atare and date in handwriting by p | ~····································· | |







# INFORMED CONSENT LEGALREPRESENTATIVE

| | STUDY TITLE: | | | |
|---|---|---|---|---|
| | | • | | ed health recommendations to the general population |
| | | | app as a strategy for gastric cancer prevention". | |
| | STUDY CODE | | 101095359 – AID | |
| | PRINCIPAL INVE | STIGATORS | To be completed | |
| | DEPARTMENT | | To be completed | |
| | CENTER | | To be completed | <u>,</u> |
| ١, _ | (Name in ha | andwriting by represents | | < <representative's and="" name="" surname="">&gt;</representative's> |
| (Name in handwriting by representative In my capacity as | | ative) | <pre>&lt;<relationship participant="" the="" to="">&gt;, of</relationship></pre> | |
| | my capacity | <u> </u> | | <pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre>&lt;<pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre></pre> |
| | (Name in ha | andwriting by representa | | |
| | | nation sheet that has | - | about the study. |
| | | stions about the stu | • | |
| | | gh information abou | | |
| I h | ave spoken to $\_\_$ | | | < <name investigator="" of="">&gt;</name> |
| | | | vriting by representativ | re) |
| | | /her participation is | • | |
| | | /she is free to withd | raw from the study | y: |
| | t any time. | | | |
| - W | /ithout giving a rea | ason. | | |
| - W | ithout this affecti | ng his/her medical o | care. | |
| I fr | eely give my conse | ent to his/her partic | ipation in the study | y. |
| I co | onsent to the use a | and processing of his | s/her personal data | a for this investigation under the conditions explained |
| in t | this information sh | neet. | • | |
| | ( C ) | | | |
| US | e of Samples | | | |
| l c | onsent to the sto | rage and use of th | e samples and ass | sociated data for this research under the conditions |
| ex | olained in this info | rmation sheet. | | |
| $\square$ Y | 'ES | NO | | |
| | | • | | nation generated from the research (genetic or non- |
| gei | netic, depending o | n the case) that ma | y be relevant and a | applicable to my health or that of my family members: |
| $\square$ Y | 'ES | NO | Contact telepho | one or email |
| | | | - | |
| I co | onsent to be conta | icted if there is a ne | ed for further infor | mation or additional biological samples. |
| $\square$ Y | 'ES | NO | Contact telepho | one or email |
| | | | · | |
| l w | ill receive a signed | d and dated copy of | this informed cons | ent form |
| | Signature of logal | representative, rela | tive or related | Investigator's Signature |
| | | representative, rela | tive of Telateu | investigator a dignature |
| | party | , | | Date: / / |
| (Sig | Date:// | <br>ndwriting by representa | tive) | Date:/ |
| 10 | | | 1 | |







# INFORMED CONSENT BEFORE WITNESSES

| STUDY CODE | | pp as a strategy for gastric cancer prevention". 101095359 – AIDA | |
|---|---|---|---|
| PRINCIPAL INV | /ESTIGATORS | To be completed | _ |
| DEPARTMENT | | To be completed | |
| CENTER | | To be completed | |
| l, | | < <witness's and="" name="" surname="">&gt;</witness's> | |
| • | nandwriting by witness) | | |
| as a witness, state t | | <pre>&lt;&lt; participant's name and surname &gt;&gt; [Name in handwriting by witness]</pre> | |
| | ( | intality in hallowitting by withessy | |
| has been inform | ed and has read the | e information sheet about the study, and therefore: | |
| He/she has read the | e information sheet | that has been given to him/her about the study. | |
| Was able to ask que | | · | |
| Has received enoug | | | |
| Has spoken to | | <pre>&lt;<name investigator="" of="">&gt;</name></pre> | |
| | · · | dwriting by witness) | |
| Understands that h | | · | |
| | e/she is free to with | hdraw from the study: | |
| - At any time. | | | |
| - Without giving a r | eason. | | |
| <ul> <li>Without this affec</li> </ul> | _ | | |
| Freely gives his/her | consent to particip | pate in the study. | |
| Freely gives his/her<br>Consents to the use | consent to participe and processing of | | d |
| Freely gives his/her | consent to participe and processing of | pate in the study. | d |
| Freely gives his/her<br>Consents to the use<br>in this information s | consent to participe and processing of | pate in the study. | d |
| Freely gives his/her<br>Consents to the use | consent to participe and processing of | pate in the study. | d |
| Freely gives his/her Consents to the use in this information successions. | consent to participe<br>and processing of<br>sheet. | pate in the study.<br>his/her personal data for this investigation under the conditions explained | |
| Freely gives his/her Consents to the use in this information successful to the Store Consent to the store consent consent to the store consent c | consent to participe and processing of sheet. | pate in the study. | |
| Freely gives his/her Consents to the use in this information: <u>Use of Samples</u> Consent to the stoexplained in this information. | consent to participe and processing of sheet. brage and use of to formation sheet. | pate in the study.<br>his/her personal data for this investigation under the conditions explained | |
| Freely gives his/her Consents to the use in this information successful to the Store Consent to the store consent consent to the store consent c | consent to participe and processing of sheet. | pate in the study.<br>his/her personal data for this investigation under the conditions explained | |
| Freely gives his/her Consents to the use in this information successive of Samples Consent to the stoe explained in this information. | consent to participe and processing of sheet. brage and use of the formation sheet. | his/her personal data for this investigation under the conditions explained his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition | าร |
| Freely gives his/her Consents to the use in this information: Use of Samples Consent to the sto explained in this information YES Would like the study | consent to participe and processing of sheet. brage and use of tormation sheet. NO NO No | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor | ns<br>n- |
| Freely gives his/her Consents to the use in this information: Use of Samples Consent to the sto explained in this information YES Would like the studgenetic, depending | consent to participe and processing of sheet. brage and use of tormation sheet. NO NO No | his/her personal data for this investigation under the conditions explained his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition | ns<br>n- |
| Freely gives his/her Consents to the use in this information subsection of the store of Samples Consent to the store explained in this information of the store of Samples Would like the store genetic, depending members: | consent to participe and processing of sheet. brage and use of the formation sheet. NO ly doctor to inform on the case) that it | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her family | ns<br>n- |
| Freely gives his/her Consents to the use in this information subsection of the store of Samples Consent to the store explained in this information of the store of Samples Would like the store genetic, depending members: | consent to participe and processing of sheet. brage and use of tormation sheet. NO NO No | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor | ns<br>n- |
| Freely gives his/her Consents to the use in this information such that in this information such that it is consent to the store explained in this information. YES Would like the study genetic, depending members: YES | consent to participe and processing of sheet. orage and use of the formation sheet. NO ly doctor to inform on the case) that in | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information subsection of the store of Samples Consent to the store explained in this information of the store explained in this information. YES Would like the store genetic, depending members: YES Consents to be consents to be consents. | consent to participe and processing of sheet. orage and use of tormation sheet. NO ly doctor to inform on the case) that in the case and the case are consequently the case are case are consequently the case are consequently | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her familicontact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information subsection of the store of Samples Consent to the store explained in this information of the store explained in this information. YES Would like the store genetic, depending members: YES Consents to be consents to be consents. | consent to participe and processing of sheet. orage and use of the formation sheet. NO ly doctor to inform on the case) that in | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information surples Use of Samples Consent to the storexplained in this information surples Would like the studgenetic, depending members: YES Consents to be consents to be consents to be consents. | consent to participe and processing of sheet. orage and use of the formation sheet. NO ly doctor to inform on the case) that in the case if there is a reconstruction. | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information surples Use of Samples Consent to the storexplained in this information surples Would like the studgenetic, depending members: YES Consents to be consents to be consents to be consents. | consent to participe and processing of sheet. orage and use of the formation sheet. NO ly doctor to inform on the case) that in the case if there is a reconstruction. | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her familicontact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information surples Use of Samples Consent to the storexplained in this information surples Would like the studgenetic, depending members: YES Consents to be consents to be consents to be consents. | consent to participe and processing of sheet. orage and use of the formation sheet. NO ly doctor to inform on the case) that in the case if there is a reconstruction. | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information surples Use of Samples Consent to the storexplained in this information surples Would like the studgenetic, depending members: YES Consents to be consents to be consents to be consents to be consents. | consent to participe and processing of sheet. brage and use of the formation sheet. NO ly doctor to inform on the case) that in the case and the case are are are and the copy of the c | his/her personal data for this investigation under the conditions explained the samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |
| Freely gives his/her Consents to the use in this information surples Use of Samples Consent to the storexplained in this information surples Would like the studgenetic, depending members: YES Consents to be consents to be consents to be consents. | consent to participe and processing of sheet. brage and use of tromation sheet. NO ly doctor to inform on the case) that in the case and the case are are and the case are are are and and dated copy on the case. | his/her personal data for this investigation under the conditions explained he samples and associated data for this research under the condition him/her about information generated from the research (genetic or nor may be relevant and applicable to his/her health or that of his/her famil Contact telephone or email | ns<br>n- |